CLINICAL TRIAL: NCT07273643
Title: Characterization of Extracellular Vesicles From the Cord Blood of Extremely Preterm New Borns and Their Correlation With Severe Morbidity and Mortality
Acronym: VEEP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM U1046 Physiologie et médecine expérimentale du coeur et des muscles (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL25_0241
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Intraventricular Hemorrhage; Pulmonary Hemorrhage; Death; ELGAN (22-28SA); Bronchopulmonary Dysplasia (BPD); Shock; Extracellular Vesicles; Enterocolitis, Necrotizing
Keywords: ELGAN; Extremely Low Gestational Age Newborn (ELGAN); Extracellular vesicles; EVs; Intraventricular hemorrage; Pulmonary hemorrhage; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Death; Bronchopulmonary Dysplasia; Shock; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Blood samples will be centrifuged to remove blood cells and obtain plasma, which will be frozen for later analysis of extracellular vesicles (EVs). These samples will be stored for at least five years. Future studies, such as microRNA analysis, functional tests, or microscopic visualization, may also be performed. All of this sample will be anonymized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extremely Low Gestational Age Newborns without severe morbidity or mortality: Extremely Low Gestational Age Newborns (ELGANs) born at Montpellier Hospital before 28 weeks of gestation, who were admitted to the neonatal unit, had cord blood collected at birth, and did not experience severe morbidity (early shock, intraventricular hemorrhage, or pulmonary hemorrhage) or death before discharge.
  Interventions: Biological: Venous Cord blood sample; Biological: Arterial cord blood sample
- Extremely Low Gestational Age Newborns with severe morbidity or mortality: Extremely Low Gestational Age Newborns (ELGANs) born at Montpellier Hospital before 28 weeks of gestation, who were admitted to the neonatal unit, had cord blood collected at birth, and experienced severe morbidity (early shock, intraventricular hemorrhage, or pulmonary hemorrhage) or death before discharge.
  Interventions: Biological: Venous Cord blood sample; Biological: Arterial cord blood sample

INTERVENTIONS:
Biological: Venous Cord blood sample — Venous cord blood sample will be collected at birth (10 mL; if not possible, a minimum of 3 mL) from the umbilical vein into an EDTA tube. Plasma was isolated from blood cells by two centrifugation steps. Extracellular vesicles (EVs) were then isolated from plasma using additional centrifugation and ultracentrifugation steps. EVs were sized and counted using a Zetasizer, and their cellular origin was characterized by nanocytometry.
  Other Names: EVs extraction and characterization; Blood centrifugation
Biological: Arterial cord blood sample — Arterial cord blood sample will be collected at birth (10 mL; if not possible, a minimum of 3 mL) from the umbilical vein into an EDTA tube for the five first inclusions (succeed). Plasma was isolated from blood cells by two centrifugation steps. Extracellular vesicles (EVs) were then isolated from plasma using additional centrifugation and ultracentrifugation steps. EVs were sized and counted using a Zetasizer, and their cellular origin was characterized by nanocytometry.
  Other Names: EVs extraction and characterization; Blood centrifugation

SUMMARY:
This study aims to understand the role of extracellular vesicles (EVs) in extremely premature infants, those born before 28 weeks of gestation. EVs are tiny particles released by cells that carry important information about the body's condition. In extremely premature infants, blood vessels may not function properly, leading to serious health problems such as bleeding in the brain, lung injury, or severe infections.

Researchers believe that analyzing EVs in the umbilical cord blood of these infants may help predict which babies are at higher risk of developing these complications. By studying the size, number, and type of EVs, the team hopes to identify early markers that can guide doctors in providing better care.

The study will collect cord blood from 30 eligible infants born at the CHU of Montpellier. Blood samples will be processed to isolate platelet-poor plasma, which contains EVs. This plasma will be stored in a biobank, allowing future research on EVs and their role in extreme prematurity. EVs will then be analyzed in the laboratory to assess their characteristics and any links to severe health issues.

The findings from this study could improve understanding of circulatory problems in extremely premature infants, help identify early predictors of severe complications, and inform better monitoring and treatment strategies. The creation of a plasma biobank also provides a valuable resource for future research to enhance care and outcomes for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Mother over 18 years old, able to speak and understand French
* Newborn less than 28 weeks of gestation, born and hospitalized at Montpellier University Hospital
* Umbilical cord venous blood collected immediately after birth (from the segment between the cord clamp and the placenta), with a volume of 10 ml (which can be reduced to 3 ml if collection is difficult) into an EDTA tube.
* Parental non-opposition to the study obtained before sample collection

Exclusion Criteria:

* Stillborn infant
* Handling failure: failure to collect the sample or start the first centrifugation more than 3 hours after birth
* General regulatory criteria: failure to obtain parental non-opposition, lack of social security coverage, individuals under legal guardianship, or participation in another ongoing research study with an active exclusion period

Ages: 0 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All live-born infants born before 28 weeks of gestation (extremely preterm) who were hospitalized at Montpellier University Hospital during the inclusion period and had cord blood collected immediately after birth.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between occurence of early severe morbidity mortality and characterization of Extracellular vesicles (EVs) | Blood collection: at birth Centrifugation: within 3 hours of collection. EV isolation and analysis: up to there month after collection. Clinical informations(occurence of early severe morbidity and mortality): through study completion, up to 1year
  The primary outcome is the correlation between occurence of early severe morbidity mortality and the characterization of Extracellular vesicles (EVs) for venous cord blood plasma :
  1. EV were isolated from venous cord blood plasma using sequential centrifugation and ultracentrifugation steps. EVs were then characterized for size (nm) and concentration (EVs/µL) using a Zetasizer, and their cellular origin was determined by nanocytometry.
  2. Early severe morbidity or mortality during the hospital stay is defined as the occurrence of at least one of the following events:
     * Refractory shock (requiring fluid resuscitation or vasopressor support)
     * Pulmonary Hemorrhage
     * Severe Intraventricular Hemorrhage (grade 3 or 4, Papille classification)
     * Death before discharge

SECONDARY OUTCOMES:
Correlation between occurrence of other morbidity before discharge and the EVs characterization | Blood collection: at birth Centrifugation: within 3 hours of collection. EV isolation and analysis: up to there month after collection. Clinical informations (occurence of other morbidity): through study completion, up to 1year.
  This secondary outcome will explore the correlation between the characterization of venous cord blood extracellular vesicles (EVs), as defined in the primary outcome, and the occurrence of other morbidities before discharge, defined as:
  * Necrotizing enterocolitis
  * Bronchopulmonary dysplasia
  * Other significant conditions
Correlation between obstetric characteristics and causes of prematurity and characterization of venous cord blood EVs. | Blood collection: at birth Centrifugation: within 3 hours of collection. EV isolation and analysis: up to there month after collection. Clinical informations (obstetric characteristics and causes of prematurity): through study completion, up to 1year
  This secondary outcome will explore the correlation between the characterization of venous cord blood extracellular vesicles (EVs), as defined in the primary outcome, and the obstetric characteristics and causes of prematurity
Comparison of Arterial and Venous Extracellular Vesicles | Blood collection: at birth Centrifugation: within 3 hours of collection. EV isolation and analysis: up to there month after collection.
  For the first five inclusions, an arterial blood sample will also be collected. Extracellular vesicles (EVs) from arterial and venous cord blood will be characterized for size, concentration, and cellular origin using the same methods as described for the primary outcome.
  Arterial and venous EV characteristics will then be compared.

REFERENCES:
- [Background] Pekarkova K, Soukup J, Kostelanska M, Sirc J, Stranak Z, Holada K. Cord Blood Extracellular Vesicles Analyzed by Flow Cytometry with Thresholding Using 405 nm or 488 nm Laser Leads to Concurrent Results. Diagnostics (Basel). 2021 Jul 22;11(8):1320. doi: 10.3390/diagnostics11081320. PMID 34441255
- [Background] Hujacova A, Brozova T, Mosko T, Kostelanska M, Stranak Z, Holada K. Platelet Extracellular Vesicles in Cord Blood of Term and Preterm Newborns Assayed by Flow Cytometry: the Effect of Delay in Sample Preparation and of Sample Freezing. Folia Biol (Praha). 2020;66(5-6):204-211. doi: 10.14712/fb2020066050204. PMID 34087976
- [Background] Galley JD, Mar P, Wang Y, Han R, Rajab A, Besner GE. Urine-derived extracellular vesicle miRNAs as possible biomarkers for and mediators of necrotizing enterocolitis: A proof of concept study. J Pediatr Surg. 2021 Nov;56(11):1966-1975. doi: 10.1016/j.jpedsurg.2021.02.016. Epub 2021 Mar 2. PMID 33785202
- [Background] Jakkula M, Le Cras TD, Gebb S, Hirth KP, Tuder RM, Voelkel NF, Abman SH. Inhibition of angiogenesis decreases alveolarization in the developing rat lung. Am J Physiol Lung Cell Mol Physiol. 2000 Sep;279(3):L600-7. doi: 10.1152/ajplung.2000.279.3.L600. PMID 10956636
- [Background] Janer J, Andersson S, Kajantie E, Lassus P. Endostatin concentration in cord plasma predicts the development of bronchopulmonary dysplasia in very low birth weight infants. Pediatrics. 2009 Apr;123(4):1142-6. doi: 10.1542/peds.2008-1339. PMID 19336373
- [Background] Baker CD, Balasubramaniam V, Mourani PM, Sontag MK, Black CP, Ryan SL, Abman SH. Cord blood angiogenic progenitor cells are decreased in bronchopulmonary dysplasia. Eur Respir J. 2012 Dec;40(6):1516-22. doi: 10.1183/09031936.00017312. Epub 2012 Apr 10. PMID 22496315
- [Background] Borghesi A, Massa M, Campanelli R, Bollani L, Tzialla C, Figar TA, Ferrari G, Bonetti E, Chiesa G, de Silvestri A, Spinillo A, Rosti V, Stronati M. Circulating endothelial progenitor cells in preterm infants with bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2009 Sep 15;180(6):540-6. doi: 10.1164/rccm.200812-1949OC. Epub 2009 Jul 2. PMID 19574444
- [Background] Zhong XQ, Yan Q, Chen ZG, Jia CH, Li XH, Liang ZY, Gu J, Wei HL, Lian CY, Zheng J, Cui QL. Umbilical Cord Blood-Derived Exosomes From Very Preterm Infants With Bronchopulmonary Dysplasia Impaired Endothelial Angiogenesis: Roles of Exosomal MicroRNAs. Front Cell Dev Biol. 2021 Mar 25;9:637248. doi: 10.3389/fcell.2021.637248. eCollection 2021. PMID 33842462
- [Background] Lal CV, Olave N, Travers C, Rezonzew G, Dolma K, Simpson A, Halloran B, Aghai Z, Das P, Sharma N, Xu X, Genschmer K, Russell D, Szul T, Yi N, Blalock JE, Gaggar A, Bhandari V, Ambalavanan N. Exosomal microRNA predicts and protects against severe bronchopulmonary dysplasia in extremely premature infants. JCI Insight. 2018 Mar 8;3(5):e93994. doi: 10.1172/jci.insight.93994. PMID 29515035
- [Background] Schiller EA, Cohen K, Lin X, El-Khawam R, Hanna N. Extracellular Vesicle-microRNAs as Diagnostic Biomarkers in Preterm Neonates. Int J Mol Sci. 2023 Jan 30;24(3):2622. doi: 10.3390/ijms24032622. PMID 36768944
- [Background] Menon R, Shahin H. Extracellular vesicles in spontaneous preterm birth. Am J Reprod Immunol. 2021 Feb;85(2):e13353. doi: 10.1111/aji.13353. Epub 2020 Oct 12. PMID 32975858
- [Background] Farrelly R, Kennedy MG, Spencer R, Forbes K. Extracellular vesicles as markers and mediators of pregnancy complications: gestational diabetes, pre-eclampsia, preterm birth and fetal growth restriction. J Physiol. 2023 Nov;601(22):4973-4988. doi: 10.1113/JP282849. Epub 2023 May 8. PMID 37070801
- [Background] Tesse A, Meziani F, David E, Carusio N, Kremer H, Schneider F, Andriantsitohaina R. Microparticles from preeclamptic women induce vascular hyporeactivity in vessels from pregnant mice through an overproduction of NO. Am J Physiol Heart Circ Physiol. 2007 Jul;293(1):H520-5. doi: 10.1152/ajpheart.01094.2006. Epub 2007 Mar 16. PMID 17369461
- [Background] Bravo MC, Lopez-Ortego P, Sanchez L, Riera J, Madero R, Cabanas F, Pellicer A. Randomized, Placebo-Controlled Trial of Dobutamine for Low Superior Vena Cava Flow in Infants. J Pediatr. 2015 Sep;167(3):572-8.e1-2. doi: 10.1016/j.jpeds.2015.05.037. Epub 2015 Jun 24. PMID 26116470
- [Background] Elsayed Y, Ahmed F. Blood pressure normative values in preterm infants during postnatal transition. Pediatr Res. 2024 Feb;95(3):698-704. doi: 10.1038/s41390-023-02788-8. Epub 2023 Sep 4. PMID 37667035
- [Background] Peeples ES, Comstock BA, Heagerty PJ, Juul SE; Preterm Erythropoietin Neuroprotection (PENUT) Trial Investigators. Blood pressure values and hypotension management in extremely preterm infants: a multi-center study. J Perinatol. 2022 Sep;42(9):1169-1175. doi: 10.1038/s41372-022-01425-2. Epub 2022 Jun 17. PMID 35715600
- [Background] McNamara PJ, Jain A, El-Khuffash A, Giesinger R, Weisz D, Freud L, Levy PT, Bhombal S, de Boode W, Leone T, Richards B, Singh Y, Acevedo JM, Simpson J, Noori S, Lai WW. Guidelines and Recommendations for Targeted Neonatal Echocardiography and Cardiac Point-of-Care Ultrasound in the Neonatal Intensive Care Unit: An Update from the American Society of Echocardiography. J Am Soc Echocardiogr. 2024 Feb;37(2):171-215. doi: 10.1016/j.echo.2023.11.016. PMID 38309835
- [Background] Singh Y, Tissot C, Fraga MV, Yousef N, Cortes RG, Lopez J, Sanchez-de-Toledo J, Brierley J, Colunga JM, Raffaj D, Da Cruz E, Durand P, Kenderessy P, Lang HJ, Nishisaki A, Kneyber MC, Tissieres P, Conlon TW, De Luca D. International evidence-based guidelines on Point of Care Ultrasound (POCUS) for critically ill neonates and children issued by the POCUS Working Group of the European Society of Paediatric and Neonatal Intensive Care (ESPNIC). Crit Care. 2020 Feb 24;24(1):65. doi: 10.1186/s13054-020-2787-9. PMID 32093763
- [Background] Conti M, Minniti M, Tine M, De Francesco M, Gaeta R, Nieri D, Semenzato U, Biondini D, Camera M, Cosio MG, Saetta M, Celi A, Bazzan E, Neri T. Extracellular Vesicles in Pulmonary Hypertension: A Dangerous Liaison? Biology (Basel). 2023 Aug 7;12(8):1099. doi: 10.3390/biology12081099. PMID 37626985
- [Background] An N, Chen Z, Zhao P, Yin W. Extracellular Vesicles in Sepsis: Pathogenic Roles, Organ Damage, and Therapeutic Implications. Int J Med Sci. 2023 Oct 16;20(13):1722-1731. doi: 10.7150/ijms.86832. eCollection 2023. PMID 37928875
- [Background] Mostefai HA, Meziani F, Mastronardi ML, Agouni A, Heymes C, Sargentini C, Asfar P, Martinez MC, Andriantsitohaina R. Circulating microparticles from patients with septic shock exert protective role in vascular function. Am J Respir Crit Care Med. 2008 Dec 1;178(11):1148-55. doi: 10.1164/rccm.200712-1835OC. Epub 2008 Aug 21. PMID 18723433
- [Background] Szatanek R, Baj-Krzyworzeka M, Zimoch J, Lekka M, Siedlar M, Baran J. The Methods of Choice for Extracellular Vesicles (EVs) Characterization. Int J Mol Sci. 2017 May 29;18(6):1153. doi: 10.3390/ijms18061153. PMID 28555055
- [Background] Thery C, Witwer KW, Aikawa E, Alcaraz MJ, Anderson JD, Andriantsitohaina R, Antoniou A, Arab T, Archer F, Atkin-Smith GK, Ayre DC, Bach JM, Bachurski D, Baharvand H, Balaj L, Baldacchino S, Bauer NN, Baxter AA, Bebawy M, Beckham C, Bedina Zavec A, Benmoussa A, Berardi AC, Bergese P, Bielska E, Blenkiron C, Bobis-Wozowicz S, Boilard E, Boireau W, Bongiovanni A, Borras FE, Bosch S, Boulanger CM, Breakefield X, Breglio AM, Brennan MA, Brigstock DR, Brisson A, Broekman ML, Bromberg JF, Bryl-Gorecka P, Buch S, Buck AH, Burger D, Busatto S, Buschmann D, Bussolati B, Buzas EI, Byrd JB, Camussi G, Carter DR, Caruso S, Chamley LW, Chang YT, Chen C, Chen S, Cheng L, Chin AR, Clayton A, Clerici SP, Cocks A, Cocucci E, Coffey RJ, Cordeiro-da-Silva A, Couch Y, Coumans FA, Coyle B, Crescitelli R, Criado MF, D'Souza-Schorey C, Das S, Datta Chaudhuri A, de Candia P, De Santana EF, De Wever O, Del Portillo HA, Demaret T, Deville S, Devitt A, Dhondt B, Di Vizio D, Dieterich LC, Dolo V, Dominguez Rubio AP, Dominici M, Dourado MR, Driedonks TA, Duarte FV, Duncan HM, Eichenberger RM, Ekstrom K, El Andaloussi S, Elie-Caille C, Erdbrugger U, Falcon-Perez JM, Fatima F, Fish JE, Flores-Bellver M, Forsonits A, Frelet-Barrand A, Fricke F, Fuhrmann G, Gabrielsson S, Gamez-Valero A, Gardiner C, Gartner K, Gaudin R, Gho YS, Giebel B, Gilbert C, Gimona M, Giusti I, Goberdhan DC, Gorgens A, Gorski SM, Greening DW, Gross JC, Gualerzi A, Gupta GN, Gustafson D, Handberg A, Haraszti RA, Harrison P, Hegyesi H, Hendrix A, Hill AF, Hochberg FH, Hoffmann KF, Holder B, Holthofer H, Hosseinkhani B, Hu G, Huang Y, Huber V, Hunt S, Ibrahim AG, Ikezu T, Inal JM, Isin M, Ivanova A, Jackson HK, Jacobsen S, Jay SM, Jayachandran M, Jenster G, Jiang L, Johnson SM, Jones JC, Jong A, Jovanovic-Talisman T, Jung S, Kalluri R, Kano SI, Kaur S, Kawamura Y, Keller ET, Khamari D, Khomyakova E, Khvorova A, Kierulf P, Kim KP, Kislinger T, Klingeborn M, Klinke DJ 2nd, Kornek M, Kosanovic MM, Kovacs AF, Kramer-Albers EM, Krasemann S, Krause M, Kurochkin IV, Kusuma GD, Kuypers S, Laitinen S, Langevin SM, Languino LR, Lannigan J, Lasser C, Laurent LC, Lavieu G, Lazaro-Ibanez E, Le Lay S, Lee MS, Lee YXF, Lemos DS, Lenassi M, Leszczynska A, Li IT, Liao K, Libregts SF, Ligeti E, Lim R, Lim SK, Line A, Linnemannstons K, Llorente A, Lombard CA, Lorenowicz MJ, Lorincz AM, Lotvall J, Lovett J, Lowry MC, Loyer X, Lu Q, Lukomska B, Lunavat TR, Maas SL, Malhi H, Marcilla A, Mariani J, Mariscal J, Martens-Uzunova ES, Martin-Jaular L, Martinez MC, Martins VR, Mathieu M, Mathivanan S, Maugeri M, McGinnis LK, McVey MJ, Meckes DG Jr, Meehan KL, Mertens I, Minciacchi VR, Moller A, Moller Jorgensen M, Morales-Kastresana A, Morhayim J, Mullier F, Muraca M, Musante L, Mussack V, Muth DC, Myburgh KH, Najrana T, Nawaz M, Nazarenko I, Nejsum P, Neri C, Neri T, Nieuwland R, Nimrichter L, Nolan JP, Nolte-'t Hoen EN, Noren Hooten N, O'Driscoll L, O'Grady T, O'Loghlen A, Ochiya T, Olivier M, Ortiz A, Ortiz LA, Osteikoetxea X, Ostergaard O, Ostrowski M, Park J, Pegtel DM, Peinado H, Perut F, Pfaffl MW, Phinney DG, Pieters BC, Pink RC, Pisetsky DS, Pogge von Strandmann E, Polakovicova I, Poon IK, Powell BH, Prada I, Pulliam L, Quesenberry P, Radeghieri A, Raffai RL, Raimondo S, Rak J, Ramirez MI, Raposo G, Rayyan MS, Regev-Rudzki N, Ricklefs FL, Robbins PD, Roberts DD, Rodrigues SC, Rohde E, Rome S, Rouschop KM, Rughetti A, Russell AE, Saa P, Sahoo S, Salas-Huenuleo E, Sanchez C, Saugstad JA, Saul MJ, Schiffelers RM, Schneider R, Schoyen TH, Scott A, Shahaj E, Sharma S, Shatnyeva O, Shekari F, Shelke GV, Shetty AK, Shiba K, Siljander PR, Silva AM, Skowronek A, Snyder OL 2nd, Soares RP, Sodar BW, Soekmadji C, Sotillo J, Stahl PD, Stoorvogel W, Stott SL, Strasser EF, Swift S, Tahara H, Tewari M, Timms K, Tiwari S, Tixeira R, Tkach M, Toh WS, Tomasini R, Torrecilhas AC, Tosar JP, Toxavidis V, Urbanelli L, Vader P, van Balkom BW, van der Grein SG, Van Deun J, van Herwijnen MJ, Van Keuren-Jensen K, van Niel G, van Royen ME, van Wijnen AJ, Vasconcelos MH, Vechetti IJ Jr, Veit TD, Vella LJ, Velot E, Verweij FJ, Vestad B, Vinas JL, Visnovitz T, Vukman KV, Wahlgren J, Watson DC, Wauben MH, Weaver A, Webber JP, Weber V, Wehman AM, Weiss DJ, Welsh JA, Wendt S, Wheelock AM, Wiener Z, Witte L, Wolfram J, Xagorari A, Xander P, Xu J, Yan X, Yanez-Mo M, Yin H, Yuana Y, Zappulli V, Zarubova J, Zekas V, Zhang JY, Zhao Z, Zheng L, Zheutlin AR, Zickler AM, Zimmermann P, Zivkovic AM, Zocco D, Zuba-Surma EK. Minimal information for studies of extracellular vesicles 2018 (MISEV2018): a position statement of the International Society for Extracellular Vesicles and update of the MISEV2014 guidelines. J Extracell Vesicles. 2018 Nov 23;7(1):1535750. doi: 10.1080/20013078.2018.1535750. eCollection 2018. PMID 30637094
- [Background] El-Khuffash AF, McNamara PJ. Neonatologist-performed functional echocardiography in the neonatal intensive care unit. Semin Fetal Neonatal Med. 2011 Feb;16(1):50-60. doi: 10.1016/j.siny.2010.05.001. Epub 2010 Jun 19. PMID 20646976
- [Background] Durrmeyer X, Marchand-Martin L, Porcher R, Gascoin G, Roze JC, Storme L, Favrais G, Ancel PY, Cambonie G; Hemodynamic EPIPAGE 2 Study Group. Abstention or intervention for isolated hypotension in the first 3 days of life in extremely preterm infants: association with short-term outcomes in the EPIPAGE 2 cohort study. Arch Dis Child Fetal Neonatal Ed. 2017 Nov;102(6):490-496. doi: 10.1136/archdischild-2016-312104. Epub 2017 Mar 16. PMID 28302697
- [Background] Rowcliff K, de Waal K, Mohamed AL, Chaudhari T. Noradrenaline in preterm infants with cardiovascular compromise. Eur J Pediatr. 2016 Dec;175(12):1967-1973. doi: 10.1007/s00431-016-2794-7. Epub 2016 Oct 15. PMID 27744568
- [Background] Paradisis M, Evans N, Kluckow M, Osborn D. Randomized trial of milrinone versus placebo for prevention of low systemic blood flow in very preterm infants. J Pediatr. 2009 Feb;154(2):189-95. doi: 10.1016/j.jpeds.2008.07.059. Epub 2008 Sep 25. PMID 18822428
- [Background] Kluckow M, Evans N. Low superior vena cava flow and intraventricular haemorrhage in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F188-94. doi: 10.1136/fn.82.3.f188. PMID 10794784
- [Background] Osborn DA, Evans N, Kluckow M. Left ventricular contractility in extremely premature infants in the first day and response to inotropes. Pediatr Res. 2007 Mar;61(3):335-40. doi: 10.1203/pdr.0b013e318030d1e1. PMID 17314693
- [Background] Rabe H, Gyte GM, Diaz-Rossello JL, Duley L. Effect of timing of umbilical cord clamping and other strategies to influence placental transfusion at preterm birth on maternal and infant outcomes. Cochrane Database Syst Rev. 2019 Sep 17;9(9):CD003248. doi: 10.1002/14651858.CD003248.pub4. PMID 31529790
- [Background] Myrhaug HT, Brurberg KG, Hov L, Markestad T. Survival and Impairment of Extremely Premature Infants: A Meta-analysis. Pediatrics. 2019 Feb;143(2):e20180933. doi: 10.1542/peds.2018-0933. PMID 30705140
- [Background] Higgins RD, Jobe AH, Koso-Thomas M, Bancalari E, Viscardi RM, Hartert TV, Ryan RM, Kallapur SG, Steinhorn RH, Konduri GG, Davis SD, Thebaud B, Clyman RI, Collaco JM, Martin CR, Woods JC, Finer NN, Raju TNK. Bronchopulmonary Dysplasia: Executive Summary of a Workshop. J Pediatr. 2018 Jun;197:300-308. doi: 10.1016/j.jpeds.2018.01.043. Epub 2018 Mar 16. No abstract available. PMID 29551318
- [Background] Gilfillan M, Bhandari A, Bhandari V. Diagnosis and management of bronchopulmonary dysplasia. BMJ. 2021 Oct 20;375:n1974. doi: 10.1136/bmj.n1974. PMID 34670756
- [Background] Bell EF, Hintz SR, Hansen NI, Bann CM, Wyckoff MH, DeMauro SB, Walsh MC, Vohr BR, Stoll BJ, Carlo WA, Van Meurs KP, Rysavy MA, Patel RM, Merhar SL, Sanchez PJ, Laptook AR, Hibbs AM, Cotten CM, D'Angio CT, Winter S, Fuller J, Das A; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Mortality, In-Hospital Morbidity, Care Practices, and 2-Year Outcomes for Extremely Preterm Infants in the US, 2013-2018. JAMA. 2022 Jan 18;327(3):248-263. doi: 10.1001/jama.2021.23580. Erratum In: JAMA. 2022 Jun 7;327(21):2151. doi: 10.1001/jama.2022.7723. PMID 35040888
- [Background] Ancel PY, Goffinet F; EPIPAGE-2 Writing Group; Kuhn P, Langer B, Matis J, Hernandorena X, Chabanier P, Joly-Pedespan L, Lecomte B, Vendittelli F, Dreyfus M, Guillois B, Burguet A, Sagot P, Sizun J, Beuchee A, Rouget F, Favreau A, Saliba E, Bednarek N, Morville P, Thiriez G, Marpeau L, Marret S, Kayem G, Durrmeyer X, Granier M, Baud O, Jarreau PH, Mitanchez D, Boileau P, Boulot P, Cambonie G, Daude H, Bedu A, Mons F, Fresson J, Vieux R, Alberge C, Arnaud C, Vayssiere C, Truffert P, Pierrat V, Subtil D, D'Ercole C, Gire C, Simeoni U, Bongain A, Sentilhes L, Roze JC, Gondry J, Leke A, Deiber M, Claris O, Picaud JC, Ego A, Debillon T, Poulichet A, Coline E, Favre A, Flechelles O, Samperiz S, Ramful D, Branger B, Benhammou V, Foix-L'Helias L, Marchand-Martin L, Kaminski M. Survival and morbidity of preterm children born at 22 through 34 weeks' gestation in France in 2011: results of the EPIPAGE-2 cohort study. JAMA Pediatr. 2015 Mar;169(3):230-8. doi: 10.1001/jamapediatrics.2014.3351. PMID 25621457
- [Background] Treluyer L, Chevallier M, Jarreau PH, Baud O, Benhammou V, Gire C, Marchand-Martin L, Marret S, Pierrat V, Ancel PY, Torchin H. Intraventricular Hemorrhage in Very Preterm Children: Mortality and Neurodevelopment at Age 5. Pediatrics. 2023 Apr 1;151(4):e2022059138. doi: 10.1542/peds.2022-059138. PMID 36919442
- [Background] Papile LA, Burstein J, Burstein R, Koffler H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr. 1978 Apr;92(4):529-34. doi: 10.1016/s0022-3476(78)80282-0. PMID 305471
- [Background] Wu TW, Noori S. Recognition and management of neonatal hemodynamic compromise. Pediatr Neonatol. 2021 Feb;62 Suppl 1:S22-S29. doi: 10.1016/j.pedneo.2020.12.007. Epub 2020 Dec 24. PMID 33485823
- [Background] Kluckow M. The Pathophysiology of Low Systemic Blood Flow in the Preterm Infant. Front Pediatr. 2018 Feb 16;6:29. doi: 10.3389/fped.2018.00029. eCollection 2018. PMID 29503814